CLINICAL TRIAL: NCT06549855
Title: PD-1 Inhibitor Combined With Progesterone Treatment in Fertility Sparing Therapy for Mismatch Repair-deficient Endometrial Cancer
Brief Title: PD-1 Inhibitor Combined With Progesterone Treatment in FST for Patients With MMRd Endometrial Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Collaborators: Peking Union Medical College Hospital (Other); Peking University Third Hospital (Other); Huazhong University of Science and Technology (Other); Tianjin Medical University (Other); Shandong University (Other); Shengjing Hospital (Other); Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Wang Jianliu, Vice-president of Peking University People's Hospital, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024MMRdECFerSp
Record Dates: First submitted 2024-07-21; First posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Endometrial Cancer; Endometrioid Carcinoma; Mismatch Repair Deficiency
Keywords: Fertility preservation; Endometrioid Carcinoma; PD-1 inhibitor
MeSH Terms: conditions — Endometrial Neoplasms; Carcinoma, Endometrioid; Turcot syndrome | interventions — sintilimab; pembrolizumab; Medroxyprogesterone Acetate; Megestrol Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD-1 Inhibitor Combined With Progesterone Treatment (Experimental): All participants
  Interventions: Drug: Sintilimab or Pembrolizumab and medroxyprogesterone acetate (MPA)/ megestrol acetate (MA)

INTERVENTIONS:
Drug: Sintilimab or Pembrolizumab and medroxyprogesterone acetate (MPA)/ megestrol acetate (MA) — 1. Sintilimab or Pembrolizumab 200mg intravenous injection, every 3 weeks
  2. MA, 320mg/MPA, 500mg, po, once a day
  Other Names: Sintilimab or Pembrolizumab and MPA/MA

SUMMARY:
The objective of this study was to investigate the feasibility of a PD-1 inhibitor in combination with progesterone as a means of preserving fertility in patients with early-stage mismatch repair-deficient (MMRd) endometrial cancer who wish to preserve fertility.

DETAILED DESCRIPTION:
Endometrial cancer (EC) is a prevalent gynecological cancer with an escalating global incidence. The standard treatment for endometrial cancer is total hysterectomy and bilateral salpingo-oophorectomy. However, given the rising incidence of endometrial cancer in younger individuals and the the delay in the age of human reproduction, the conservation of endometrial cancer has garnered heightened attention. Clinical practice has demonstrated that high-dose progesterone can reverse the lesioned endometrium, thereby providing a rationale for the conservative treatment of early-stage endometrial cancer.

PD-1 inhibitor has been utilized as a salvage treatment in many cancers including ovarian cancer, cervical cancer, lung cancer, gastric cancer and endometrial cancer. As endometrial cancer showed MMRd rates, it is assumed to be highly responsive to PD-1 inhibitor treatment. Previous literature has reported that the efficacy of progesterone therapy is limited in patients with a MMRd status.Here we want to investigate the feasibility of PD-1 inhibitor combined with progesterone in early stage endometrial cancer patients who want to preserve fertility.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 18-45 years old;
* Stage IA (FIGO 2009) ;
* Confirmed diagnosis of endometrial adenocarcinoma G1-G2 based upon D&C or hysteroscopy;
* Molecular classification of MMRd, determined by immunohistochemical (IHC) for MMR proteins and by the second generation sequencing (NGS) or microsatellite polymerase chain reaction (PCR);
* With a strong desire for fertility preservation;
* Sign the informed consent.

Exclusion Criteria:

* Stage IB(FIGO 2009) and above；
* Tumour differentiation of G3 or non-endometrioid adenocarcinoma；
* Complicated with any other malignancy；
* Contraindicated to conservative treatment or the use of pharmaceuticals.
* Contraindications to pregnancy, or judged by the researcher to be unfit for pregnancy or delivery.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 10 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2029-07 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Complete remission (CR) rate | From start of treatment to trial completion, an average of 3 months
  No endometrioid carcinoma or any proliferative lesion is found by pathology; imaging examination shows no evidence of a tumor
Time to CR | From start of treatment to trial completion, an average of 3 months
  Time to CR was calculated from the commencement of fertility-preserving treatment to the date of the initial hysteroscopic examination to confirm CR

SECONDARY OUTCOMES:
Recurrence rate | 6 months, 1 year, 2 year, 3 year, 4 year, 5 year after CR
  After complete remission, there is evidence of recurrence in pathology, and the imaging examination shows that the lesion recurrences.
Pregnancy rate | 1 year after CR
  A pregnancy test shows pregnancy after CR.
Live birth rate | 1 year after pregnancy
  The live birth rate is defined as the ratio of live births to pregnancies.
Pathological biomarker | From the start of treatment to CR，including 3 months, 6 months, 9 months, and so forth.
  pathological markers(such as Ki-67, estrogen receptor, progesterone receptor, p53, PTEN, MLH1, PMS2, MSH2, and MSH6) at each hysteroscopy
CA125 | From the start of treatment to trial completion，including 3 months, 6 months, 9 months, and so forth.
  Used as a tumor marker for disease monitoring
Adverse reactions | From the start of treatment to trial completion，including 3 months, 6 months, 9 months, and so forth.
  Any unfavorable response resulting from the administration of any pharmaceutical agent utilized as part of the therapeutic regimen.

CONTACTS AND LOCATIONS:
Overall Officials: Jianliu Wang, Professor, Study Chair — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No